CLINICAL TRIAL: NCT05503511
Title: A Single-center, Randomized, Placebo Controlled, Double-blind, Ascending Single-dose and Repeated-dose Trial to Determine the Safety and Pharmacokinetic Profile of NPT 2042 Soft-Gelatin Capsules Administered Orally to Healthy Adult Subjects
Brief Title: Safety and Pharmacokinetic Study of NPT 2042 Soft-gelatin Capsules Administered Orally to Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroPro Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NPT 2042 CL-101
Record Dates: First submitted 2022-07-28; First posted 2022-08-16 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-04

CONDITIONS: Epilepsy; Alzheimer Disease; Epilepsy Intractable
Keywords: CNS Disorder; Seizure Disorder
MeSH Terms: conditions — Epilepsy; Alzheimer Disease; Drug Resistant Epilepsy; Central Nervous System Diseases | interventions — Bumetanide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A; Cohort 1 (Experimental): QD dosing of 10mg (1 day)
  Interventions: Drug: NPT 2042 (bumetanide analog) or Matching Placebo
- Part A; Cohort 2 (Experimental): QD dosing of 50mg (1 day)
  Interventions: Drug: NPT 2042 (bumetanide analog) or Matching Placebo
- Part A; Cohort 3 (Experimental): QD dosing of 160mg (1 day)
  Interventions: Drug: NPT 2042 (bumetanide analog) or Matching Placebo
- Part B; Cohort 1 (Experimental): Every 12-hour dosing of 20mg (7 days)
  Interventions: Drug: NPT 2042 (bumetanide analog) or Matching Placebo
- Part B; Cohort 2 (Experimental): Every 12-hour dosing of 40mg (7 days)
  Interventions: Drug: NPT 2042 (bumetanide analog) or Matching Placebo
- Part B; Cohort 3 (Experimental): Every 12-hour dosing of 80mg (7 days)
  Interventions: Drug: NPT 2042 (bumetanide analog) or Matching Placebo

INTERVENTIONS:
Drug: NPT 2042 (bumetanide analog) or Matching Placebo — Soft gelatin capsules

SUMMARY:
Study NPT 2042 CL 101 is a first in human (FIH) study to evaluate the safety and pharmacokinetics (PK) of single and repeated ascending doses of NPT 2042 in healthy adult male and female subjects.

DETAILED DESCRIPTION:
The long-term goal of this program is to develop NPT 2042 an adjunct antiseizure treatment for patients with medically intractable epilepsy. Prior to evaluating efficacy in the intended patient population, safety and pharmacokinetics of NPT 2042 will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index (BMI) of 18 to 32 kg/m2, inclusive
2. A minimum body weight of 50 kg for males and 45 kg for females
3. All females must have a negative serum pregnancy test at Screening and a negative serum pregnancy test upon admission to the clinical research center.
4. Females must be of nonchild-bearing potential defined as permanently sterile (i.e., due to hysterectomy) or postmenopausal (defined as more than one year since last menstrual period).
5. Male subjects with female partners of reproductive potential must agree to practice abstinence or to use a condom (male subjects) plus an additional barrier method (female partner) of contraception for the duration of the study and for at least 90 days after dosing; subjects must also agree to refrain from sperm donation for at least 90 days after their last dose of IP.
6. Able to swallow capsules.

Exclusion Criteria:

1. Presence of active or recurring clinically-significant cardiovascular, pulmonary, renal, endocrine, hepatic, neurologic, psychiatric, immunologic, hematologic, gastrointestinal, or metabolic disease requiring medical treatment.
2. Presence of an active malignancy or a malignancy of any type within the past five years, other than squamous cell or basal cell carcinoma of the skin.
3. Personal or family history of long QT syndrome.
4. History or evidence of adverse symptoms associated with phlebotomy or blood donation (e.g., prolonged bleeding after injury or shaving, frequent epistaxis or gingival bleeding, bruises easily).
5. History of clinically significant vertigo, dizziness or orthostatic hypotension or any vasovagal syncope or recurrent presyncope in connection with orthostatic challenge.
6. Reported use of or inability to refrain from or anticipated use of during the study

   * any prescription drug within 14 days prior to dosing;
   * any nonprescription drug, nutritional supplement, or vitamin within 7 days prior to dosing; NOTE: acetaminophen is allowed at a dose of ≤2000 mg/day
   * any known enzyme-inducer or enzyme-inhibitor including St. John's Wort within 28 days prior to dosing, or
   * reported chronic exposure to enzyme inducers such as paint solvents or pesticides within 30 days of dosing.
7. Supine blood pressure (BP) less than 80/50 mmHg or greater than 140/90 mmHg.
8. Supine heart rate <40 bpm and >90 bpm.
9. History of drug abuse or current use of drugs of abuse or excessive ethanol intake
10. Current Smoking, vaping, hookah, chewing tobacco, or history of smoking/vaping/chewing any substance
11. Average consumption of ≥3 caffeine-containing beverages or xanthine-containing foods per day.
12. Positive urine drug, alcohol, or cotinine result at screening

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-20 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 11 days
  Absolute values and change from baseline after a single dose or after 7 days of repeated dosing.
Number of participants with abnormal lab test results | Up to 11 days
  Absolute values and change from baseline after a single dose or after 7 days of repeated dosing in clinical chemistry, hematology, and urinalysis.
Number of participants with abnormal vital signs | Up to 11 days
  Absolute values and change from baseline after a single dose or after 7 days of repeated dosing in vital signs (oral body temperature, respiratory rate, blood pressure, and heart rate).
Number of participants with abnormal ECG | Up to 7 days
  Absolute values and change from baseline after a single dose or after 7 days of ECG intervals.

SECONDARY OUTCOMES:
Pharmacokinetic Cmax | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Maximum (peak) observed concentration of NPT 2042.
Pharmacokinetic Tmax | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Time to maximum observed concentrations of NPT 2042.
Pharmacokinetic half-life (t1/2) | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Time to terminal elimination half-life concentrations of NPT 2042.
Pharmacokinetic AUClast | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Area under the concentration-time curve from zero to the last concentration quantifiable for NPT 2042.
Pharmacokinetic AUCinf | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Area under the plasma concentration-time curve from time zero extrapolated to infinity for NPT 2042.
Pharmacokinetic CL/F | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Apparent total plasma clearance after oral administration of NPT 2042.
Pharmacokinetic VzF | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Apparent volume of distribution during terminal elimination phase after oral administration of NPT 2042.
Dose proportionality | 0 (predose) and 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12, 24, 30, and 36 hours postdose
  Dose proportionality of NPT 2042 will be assessed using the power model.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States